CLINICAL TRIAL: NCT00704535
Title: Post-marketing Surveillance of the Safety, Tolerability and Efficacy of Ezetimibe Among Filipino Patients
Brief Title: Evaluation of the Safety, Tolerability and Efficacy of Ezetimibe on a Select Population of Filipinos With Hypercholesterolemia (Study P04748)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P04748
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2009-07-14 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Primary Hypercholesterolemia; Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with hypercholesterolemia: Subjects with hypercholesterolemia that are using Ezetimibe either alone or in combination with a statin
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — 1 tablet of 10 mg once daily
  Other Names: SCH 58235

SUMMARY:
The purpose of this study is to evaluate the overall safety, tolerability, and efficacy of Ezetimibe when used alone or in combination with a statin in patients with hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men or women, age 18 years and above.
* Patients with primary (heterozygous familial and non-familial) hypercholesterolemia or homozygous familial hypercholesterolemia.

Exclusion Criteria:

* Known hypersensitivity to Ezetimibe.
* Moderate to severe hepatic insufficiency.
* Persistent elevation of serum transaminase levels of more than 1.5 times the upper limit of normal.
* Pregnancy or lactation.
* Concomitant intake of bile acid sequestrants (resins), nicotinic acid (niacin), fibric acid (fibrates), or cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino subjects with hypercholesterolemia
Sampling Method: Probability Sample
Enrollment: 4105 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe as Prescribed by the Physician in Normal Practice: Filipino subjects with hypercholesterolemia who are using ezetimibe either alone or in combination with a statin
Period: Overall Study
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Started | 4105
Completed | 3959
Not Completed | 146
Not completed — Adverse Event | 2
Not completed — Death | 2
Not completed — Lost to Follow-up | 8
Not completed — Protocol Violation | 10
Not completed — Completed status not on Case Report Form | 124

BASELINE CHARACTERISTICS:
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was not reported for 10 subjects
  years | 54.62 (11.60)
Sex/Gender, Customized [Number; unit: participants] — Gender was not reported for 13 subjects
  participants
    Female | 2175
    Male | 1930

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Number of Subjects With at Least One Adverse Event
Description: Evaluation of the overall safety of ezetimibe as measured by number of subjects who experienced at least one adverse event
Time Frame: 28 days after Visit 1
Measure: Number; unit: subjects
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
subjects | 45

2. Secondary Outcome: To Evaluate the Efficacy of Ezetimibe in Lowering Serum Cholesterol Levels 28 Days After Visit 1 (Baseline)
Description: Change in mean total cholesterol values
Time Frame: 28 days after Visit 1
Population: All enrolled subjects who had both baseline and post-treatment samples collected for cholesterol measurements
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4083
mg/dL | -62.70 (47.05)

3. Primary Outcome: Safety as Measured by Number and Type of Adverse Events.
Description: Evaluation of the overall safety of ezetimibe as measured by the number and type of adverse events.
Time Frame: 28 days after Visit 1
Measure: Number; unit: adverse events
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
adverse events
  gastrointestinal upset | 2
  abdominal pain | 4
  body weakness | 1
  constipation | 3
  crampy abdominal pain | 1
  diarrhea | 6
  dizziness | 4
  epigastric discomfort | 1
  flatulence | 2
  headache | 13
  leg cramps/muscle pain | 1
  mild myalgia | 2
  myalgia | 4
  nausea | 7
  oily flatus | 1
  urticaria | 1
  vague abdominal discomfort | 1

4. Primary Outcome: Safety as Measured by Severity of Adverse Events as Determined by the Investigator
Description: To evaulate the safety of ezetimibe as measured by severity of adverse events, as determined by the investigator
Time Frame: 28 days after Visit 1
Measure: Number; unit: adverse events
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
adverse events
  Mild adverse events | 49
  Moderate adverse events | 4
  Severe adverse events | 1

5. Primary Outcome: Safety as Measured by Adverse Event Relatedness to Study Drug as Reported by the Investigator.
Description: To evaluate the overall safety of ezetimibe as measured by adverse event relatedness to study drug as reported by the investigator.
Time Frame: 28 days after Visit 1
Measure: Number; unit: adverse events
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
adverse events
  Related to treatment | 20
  Not related to treatment | 8
  Relatedness not reported | 26

6. Primary Outcome: Safety as Measured by Dose Adjustment Upon Incidence of an Adverse Event
Description: To evaluate the overall safety of ezetimibe as measured by action taken by the investigator upon incidence of an adverse event
Time Frame: 28 days after Visit 1
Measure: Number; unit: adverse event
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
adverse event
  Treatment dosage unchanged | 45
  Treatment dosage reduced | 6
  Treatment temporarily discontinued | 3

7. Primary Outcome: Safety as Measured by Outcome of Adverse Events
Description: To evaluate overall safety of ezetimibe as measured by outcome of adverse events
Time Frame: 28 days after Visit 1
Measure: Number; unit: adverse events
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
adverse events
  Adverse event cleared | 49
  Adverse event still present | 2
  Adverse event outcome not reported | 3

8. Primary Outcome: Tolerability as Measured by Subject Self-assessment
Description: Evaluation of the overall tolerability of ezetimibe as measured by subject self-assessment
Time Frame: 28 days after Visit 1
Measure: Number; unit: subjects
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Number analyzed (Participants) | 4105
subjects
  Excellent | 1325
  Very good | 1956
  Good | 713
  Fair | 54
  Poor | 3
  Not reported | 54

ADVERSE EVENTS:
Arm/Group | Ezetimibe as Prescribed by the Physician in Normal Practice
Serious Adverse Events (participants affected / at risk) | 3/4105
Other Adverse Events (participants affected / at risk) | 0/4105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe as Prescribed by the Physician in Normal Practice (N=4105)
Sepsis (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The prescribing physicians and investigators of this trial will not publish the results of any part of the study without previous written authorization from the sponsor.